CLINICAL TRIAL: NCT06855810
Title: Chinese Children's Cancer Group T-cell Acute Lymphoblastic Leukemia -2025 Project
Brief Title: Newly-diagnosed Pediatric T-cell ALL Protocol
Acronym: CCCG-TALL-2025
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IIT2025014
Record Dates: First submitted 2025-02-04; First posted 2025-03-04 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Acute Lymphoblastic Leukemia; Childhood Leukemia, Acute Lymphoblastic; T Cell Acute Lymphoblastic Leukemia/Lymphoblastic Lymphoma
Keywords: dasatinib; venetoclax; homoharringtonine
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma | interventions — venetoclax; Asparaginase; Vincristine; Cytarabine; Methotrexate; Daunorubicin; Dexamethasone; Dasatinib; Homoharringtonine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- (near)ETP-ALL (Experimental): All T-ALL patients will receive 8 mg/m2/day dexamethasone in induction therapy. For all ETP/near-ETP T-ALL patients, venetoclax will replace daunorubicin in induction therapy. CAT will replace CAT+ during early intensification. Venetoclax will replace daunorubicin in interim therapy 2 and 4. In maintenance therapy 2, the CTX+Ara-C treatment cycles are reduced to 5, in order to minimize the impact of alkylating agents on fertility.
  Interventions: Drug: Venetoclax
- nonETP-TALL-Das Group (Experimental): All T-ALL patients will receive 8 mg/m2/day dexamethasone in induction therapy. All non-ETP T-ALL patients will receive dasatinib after initial window phase in induction therapy. For non-ETP T-ALL patients with MRD <0.01% on day 46, CAT will replace CAT+ during early intensification, and patients will be continuously subjected to dasatinib combined with chemotherapy during early intensification, interim tharapy, reinduction therapy and maintenance therapy. In maintenance therapy 2, the CTX+Ara-C treatment cycles are reduced to 5, in order to minimize the impact of alkylating agents on fertility.
  Interventions: Drug: Dasatinib
- nonETP-TALL-HHT Group (Experimental): All T-ALL patients will receive 8 mg/m2/day dexamethasone in induction therapy. All non-ETP T-ALL patients will receive dasatinib after initial window phase in induction therapy. For non-ETP T-ALL patients with MRD ≥0.01% on day 46，CAT+ will be replaced with randomized doses of homoharringtonine (HHT) during early intensification, and HHT will be administrated during reinduction therapy. In maintenance therapy 2, the CTX+Ara-C treatment cycles are reduced to 5, in order to minimize the impact of alkylating agents on fertility.
  Interventions: Drug: homoharringtonine

INTERVENTIONS:
Drug: Venetoclax — All T-ALL patients will receive 8 mg/m2/day dexamethasone in induction therapy. For all ETP/near-ETP T-ALL patients, venetoclax will replace daunorubicin in induction therapy. CAT will replace CAT+ during early intensification. Venetoclax will replace daunorubicin in interim therapy 2 and 4. In maintenance therapy 2, the CTX+Ara-C treatment cycles are reduced to 5, in order to minimize the impact of alkylating agents on fertility.
  Other Names: Asparaginase; Vincristine; Cyclophosphomide; Cytarabine; 6-MP; Methotrexate; Daunorubicin; Dexamethasone
  Arms: (near)ETP-ALL
Drug: Dasatinib — All T-ALL patients will receive 8 mg/m2/day dexamethasone in induction therapy. All non-ETP T-ALL patients will receive dasatinib after initial window phase in induction therapy. For non-ETP T-ALL patients with MRD <0.01% on day 46, CAT will replace CAT+ during early intensification, and patients will be continuously subjected to dasatinib combined with chemotherapy during early intensification, interim tharapy, reinduction therapy and maintenance therapy. In maintenance therapy 2, the CTX+Ara-C treatment cycles are reduced to 5, in order to minimize the impact of alkylating agents on fertility.
  Other Names: Dexamethasone; Asparaginase; Vincristine; Daunorubicin; Cyclophosphomide; Cytarabine; 6-MP; Methotrexate
  Arms: nonETP-TALL-Das Group
Drug: homoharringtonine — All T-ALL patients will receive 8 mg/m2/day dexamethasone in induction therapy. All non-ETP T-ALL patients will receive dasatinib after initial window phase in induction therapy. For non-ETP T-ALL patients with MRD ≥0.01% on day 46，CAT+ will be replaced with randomized doses of homoharringtonine (HHT) during early intensification, and HHT will be administrated during reinduction therapy. In maintenance therapy 2, the CTX+Ara-C treatment cycles are reduced to 5, in order to minimize the impact of alkylating agents on fertility.
  Other Names: Dexamethasone; Asparaginase; Vincristine; Daunorubicin; Cyclophosphomide; Cytarabine; 6-MP; Methotrexate
  Arms: nonETP-TALL-HHT Group

SUMMARY:
This is a prospective, multicenter study conducted within the Chinese Children's Cancer Group (CCCG). The study aims to evaluate whether the addition of three novel agents, dasatinib, venetoclax and homoharringtonine, can improve the minimal residual disease (MRD)-negative remission rate, enhance event-free survival (EFS), and reduce the cumulative incidence of relapse (CIR) in pediatric patients with newly diagnosed T-cell acute lymphoblastic leukemia (T-ALL).

DETAILED DESCRIPTION:
The CCCG-T-ALL-2025 protocol will be modified as following based on the above analysis of the CCCG-ALL-2020 protocol.

1. All T-ALL patients will receive 8 mg/m2/day dexamethasone in induction therapy.
2. All non-ETP T-ALL patients will receive dasatinib after initial window phase in induction therapy.
3. non-ETP T-ALL patients with MRD ≥ 0.01% on day 46 will be stratified and randomized to receive different doses of homoharringtonine during early intensification.
4. For all ETP/near-ETP T-ALL patients, venetoclax will replace daunorubicin in induction therapy.
5. For all ETP/near-ETP T-ALL patients, venetoclax will replace daunorubicin in interim therapy 2 and 4.
6. CAT will replace CAT+ during early intensification, and will be administrated to all ETP/near-ETP patients, as well as non-ETP patients with MRD< 0.01% on day 46.

2.11.7 In maintenance therapy 2, the CTX+Ara-C treatment cycles are reduced to 5, in order to minimize the impact of alkylating agents on fertility.

2.11.8 Add drug sensitivity testing for T-ALL.

ELIGIBILITY:
Inclusion Criteria:

1. Age older than 1 month to younger than 18 years.
2. Diagnosis of acute lymphoblastic leukemia by bone marrow morphology.
3. Diagnosis of T-ALL by immunophenotyping.

Exclusion Criteria:

1. B-ALL
2. AML
3. Acute leukemias of ambiguous lineage diagnosed according to WHO or EGIL criteria.
4. ALL evolved from chronic myeloid leukemia (CML).
5. Down's syndrome, or major congenital or hereditary disease with organ dysfunction
6. Secondary leukemia
7. Known underlying congenital immunodeficiency or metabolic disease
8. Congenital heart disease with cardiac insufficiency.
9. Treated with glucocorticoids for ≥14 days, or ABL kinase inhibitors for > 7 days within one month before enrollment, or any chemotherapy or radiotherapy within 3 months before enrollment (except for emergency radiotherapy to relieve airway compression)
10. Any significant comorbidities or psychiatric disorders that may impact patient safety, compliance, informed consent, study participation, follow-up, or the interpretation of study results. In such cases, all participating sites must report directly to the PI to determine whether the patient meets exclusion criteria.
11. Severe malnutrition, active infections, heart failure, or chemotherapy intolerance.

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 610 (Estimated)
Dates: Start 2025-03-11 (Actual); Primary Completion 2030-06 (Estimated); Study Completion 2031-06 (Estimated)

PRIMARY OUTCOMES:
End-of-induction(EOI) measurable residual diseases (MRD)-negativity rate in patients with non-ETP T-ALL treated with dasatinib plus 4-drug induction compared to those treated with 4-drug induction in CCCG-ALL-2020 | The expected study duration is approximately 5 years.
  For this objective a one-sided comparison of probabilities (proportions) will be made. Let p1 and p2 be the probability of aciieving negative EOI MRD on the CCCG-ALL-2020 (historical control) and the current study respectively, then the one-sided alternative hypothesis H0: p2=p1 vs. H1: p2>p1 will be tested. The procedure of two-sample comparison of proportions with the Z-statistic (Normal approximation) will be applied.
  The current CCCG-ALL2020 data show that among 573 evaluable patients 510 (89%) achaived negative EOI MRD. Benchmarking on these as historical data, a total sample size of n=550 and interim sample size n1=300 provides sufficient popwer for the planned analyses outlined above if the true MRD negativity probability is 0.92 or higher, as shown in the table below.
  An interim analysis at n1=300 evaluable patients will be conducted for possible abstract submission or publication.
For non-ETP T-ALL patients with positive measurable residual diseases (MRD) on day 46, to compare MRD-negativity rate before consolidation between those receiving single agent homoharringtonine at dose of 1mg/m2 vs. 2mg/m2 for 7 days | The expected study duration is approximately 5 years.
  The comparison will be condicted by testing the two-sided hypothesis H0: p1=p2 vs. H1: p1≠p2, using the Z test (normal approximation) at alpha=0.10 level.
  The investigators anticipate approximately 40 patients available to be randomized. The participants will be randomized at 1:1 ratio into the two treatment arms, with 20 patients per arm. Stratified block-wise randomization will be applied with block size of 4. The randomization will be stratified by the EOI MRD level as <1% and >=1%.
End of induction (EOI) measurable residual diseases (MRD)-negativity rate with venetoclax plus 3-drug induction, compared to those treated with 4-drug induction on CCCG-ALL-2020 in treating ETP/near-ETP T-ALL. | The expected study duration is approximately 5 years.
  The investigators anticipate at least 60 evaluable ETP participants. The analysis will be conducted by testing H0: p2=p1 vs. H1: p2>p1, where p1, p2 are MRD-negative probabilities in the CCCG-ALL-2020 and the current study respectively. The Z-statistic (normal approximation) based procedure will be applied.
In interim therapies 2 and 4, venetoclax replaced daunorubicin to evaluate whether this change could improve event-free survival compared to similar patients on CCCG-ALL-2020 in treating ETP/near-ETP T-ALL. | The expected study duration is approximately 5 years.
  The investigators anticipate at least 60 evaluable participants. The event-free survival function will be estimated by the Kaplan-Meier method. Comparison will be conducted using the two-sided log-rank test.

SECONDARY OUTCOMES:
Event-free survival (EFS) of patients treated with this therapy, in comparison to historical regimens. | Approximately 6.5 years.
  The EFS functions will be estimated by the Kaplan-Meier method along with 95% confidence intervals at specified timepoints (e.g., 1, 3, 5 years since diagnosis). Standard error will be estimated using the default procedure in R. Follow up of the historical comparison cohort (CCCG-ALL-2020 and 2015) will continue during the course of the current trial. Comparisons of EFS will be performed using two-sided log-rank test. Multivariable regression modeling including trial (CCCGALL-2025 vs. 2020 or 2015) and other known prognostic factors as main effects may also be performed, using the Cox models.
Overall survival (OS) of patients treated with this therapy, in comparison to historical regimens | Approximately 6.5 years.
  The OS functions will be estimated by the Kaplan-Meier method along with 95% confidence intervals at specified timepoints (e.g., 1, 3, 5 years since diagnosis). Comparison of OS functions will be conducted using the two-sided log-rank test. Standard error will be estimated using the default procedure in R. Follow up of the historical comparison cohort (CCCG-ALL-2020 and 2015) will continue during the course of the current trial. Comparisons of OS will be performed using two-sided log-rank test. Multivariable regression modeling including trial (CCCGALL-2025 vs. 2020 or 2015) and other known prognostic factors as main effects may also be performed, using the Cox models.
Cumulative incidence of relapse (CIR) of this therapy, in comparison to historical regimens. | Approximately 6.5 years.
  CIR functions of relapse will be estimated by the Kalbafleisch-Prentice method. Follow up of the historical comparison cohort (CCCG-ALL-2020 and 2015) will continue during the course of the current trial. Comparisons of CIR will be performed by Gray's test. Multivariable regression modeling including trial (CCCGALL-2025 vs. 2020 or 2015) and other known prognostic factors as main effects may also be performed, using the Fine-Gray models.
Incidence of Grade 4 Treatment-Emergent Adverse Events (TEAE) associated with venetoclax and homoharringtonine | Up to 30 days after last dose of study treatment
  Proportions of grade-4 TEAEs in each treatment phase will be estimated by the sample proportions along with exact 95% confidence intervals. Cumulative incidences of various grade-3 or higher AEs throughout therapy will be estimated by the Kalbafleisch-Prentice method; death, relapse and other events rendering off therapy before completion are regarded as competing risks.

OTHER OUTCOMES:
To explore the pharmacokinetic profiles of bioavailability for homoharringtonine and venetoclax with Peak Plasma Concentration (Cmax) | Up to 30 days after last dose of study drug administration
  To interpret drug bioavailability, Peak Plasma Concentration (Cmax) will be calculated to qualifies the maximum exposure of the body to the drug overtime . Descriptive statistics (e.g., mean, standard deviation, five-number summary) are used to summarize the data, while visualizations like box plots and line graphs are employed to depict the drug's behavior in the body. It is recommended that centers with the appropriate resources and interest consider undertaking these studies.
To explore the pharmacokinetic profiles of bioavailability for homoharringtonine and venetoclax with Area Under the Plasma Concentration-Time Curve (AUC) | Up to 30 days after last dose of study drug administration
  To interpret drug bioavailability, Area Under the Plasma Concentration-Time Curve (AUC) will be calculated to qualifies the total exposure of the body to the drug overtime . Descriptive statistics (e.g., mean, standard deviation, five-number summary) are used to summarize the data, while visualizations like box plots and line graphs are employed to depict the drug's behavior in the body. It is recommended that centers with the appropriate resources and interest consider undertaking these studies.
To explore the pharmacokinetic profiles of absorbance duration for homoharringtonine and venetoclax with Time to Peak Concentration (Tmax) | Up to 30 days after last dose of study drug administration
  To understand how soon of drug absorbance duration, Time to Peak Concentration (Tmax) will be analyzed. Comprehensive descriptive statistics (e.g., mean, standard deviation, five-number summary) are used to summarize the data, while visualizations like box plots and line graphs are employed to depict the drug's behavior in the body. It is recommended that centers with the appropriate resources and interest consider undertaking these studies.
To explore the pharmacokinetic profiles of absorbance duration for homoharringtonine and venetoclax with Clearance (Cl) | Up to 30 days after last dose of study drug administration
  To understand how efficiently the body eliminates the drug , Clearance (CI) will be analyzed to calculate the volume of plasma from which the drug is completely removed per unit of time. Comprehensive descriptive statistics (e.g., mean, standard deviation, five-number summary) are used to summarize the data, while visualizations like box plots and line graphs are employed to depict the drug's behavior in the body. It is recommended that centers with the appropriate resources and interest consider undertaking these studies.
To explore the pharmacodynamic profiles of homoharringtonine and venetoclax. | Up to 30 days after last dose of study drug administration
  To outline the therapeutic effects from pharmarcotyping experiments, parameters as EC50 (the concentration of drug at which 50% of the maximal effect is observed) will be calculated from the dose-response curve. Visualizations as dose-response curves and concentration-effect curves are employed to depict the drug's efficacy against concentration. It is recommended that centers with the appropriate resources and interest consider undertaking these studies.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaofan Zhu, MD, Principal Investigator — Institute of Hematology and Blood Diseases Hospital, CAMS & PUMC
Locations (27):
- China (26):
  - Anhui Medical University Second Affiliated Hospital, Hefei, Anhui
  - Anhui Provincial Children's Hospital, Hefei, Anhui
  - Chongqing Medical University Affiliated Children's Hospital, Chongqing, Chongqing Municipality
  - Fujian Medical University Union Hospital, Fuzhou, Fujian
  - Guangzhou Women and Children's Medical Center, Guangzhou, Guangdong
  - Nanfang Hospital, Southern Medical University, Guangzhou, Guangdong
  - The People's Hospital of Guangxi Zhuang Autonomous Region, Nanning, Guangxi
  - The Affiliated Hospital of Guizhou Medical University, Guiyang, Guizhou
  - Tongji Hospital of Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - Union Hospital of Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - Wuhan Children's Hospital, Wuhan, Hubei
  - Hunan Children's Hospital, Changsha, Hunan
  - The Third Xiangya Hospital of the Central South University, Changsha, Hunan
  - Xiangya Hospital Central South University, Changsha, Hunan
  - Nanjing Children's Hospital Affiliated to Nanjing Medical University, Nanjin, Jiangsu
  - Children's Hospital of Soochow University, Suzhou, Jiangsu
  - Jiangxi Provincial Children's Hospital, Nanchang, Jiangxi
  - Qilu Hospital of Shandong University, Jinan, Shandong
  - Affiliated Hospital of Qingdao University, Qingdao, Shandong
  - Children's Hospital of Fudan University, Shanghai, Shanghai Municipality
  - Shanghai Children's Hospital, Shanghai, Shanghai Municipality
  - Shanghai Children's Medical Cener, Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality
  - Xi'an Northwest Women and Children Hospital, Xi’an, Shanxi
  - Shenzhen Children's Hospital, Shenzhen, Shenzhen
  - West China Second University Hospital, Chengdu, Sichuan
  - Institute of Hematology and Blood Diseases Hospital, CAMS & PUMC, Tianjin, Tianjin Municipality
- Hong Kong Children's Hospital, Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Yes
1. Demographic Data: Age, sex, and other relevant baseline characteristics.
  2. Treatment Information: Data on interventions received by participants, including dosage, treatment cycles, and duration.
  3. Outcome Measures: Detailed information on primary and secondary outcome measures, such as response rates, survival rates, adverse events, and any the pre-specified endpoints.
  4. Adverse Events: Data on all reported adverse events, including severity, duration, and outcome.
  5. Laboratory Data: Results from laboratory tests, such as blood counts, biochemical markers, or molecular analysis.
  6. Medical History: Pre-existing conditions, comorbidities, and prior treatments or interventions.
  7. Vital Signs: relevant physiological data.
  8. Efficacy and Safety Data: Any data relating to the efficacy (e.g., event-free survival) and safety (e.g., adverse effects) of the treatment.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: IPD will be made available upon publication of the primary trial results or after trial completion, whichever occurs first, starting on 2032, and will remain accessible for 5 years.
Access Criteria: Researchers, healthcare professionals who meet the criteria for access (e.g., academic researchers conducting secondary analyses or regulatory bodies reviewing safety data) will be able to request access to de-identified IPD and supporting information. Access will be facilitated through clinical trials.gov/emailing to PI, where users can submit a request and provide a research proposal. Data access will be granted after a formal review and approval process, subject to compliance with the data-sharing agreement and confidentiality terms.
URL: http://cccg.nipher.com/cccg/

REFERENCES:
- [Background] Teachey DT, Devidas M, Wood BL, Chen Z, Hayashi RJ, Hermiston ML, Annett RD, Archer JH, Asselin BL, August KJ, Cho SY, Dunsmore KP, Fisher BT, Freedman JL, Galardy PJ, Harker-Murray P, Horton TM, Jaju AI, Lam A, Messinger YH, Miles RR, Okada M, Patel SI, Schafer ES, Schechter T, Singh N, Steele AC, Sulis ML, Vargas SL, Winter SS, Wood C, Zweidler-McKay P, Bollard CM, Loh ML, Hunger SP, Raetz EA. Children's Oncology Group Trial AALL1231: A Phase III Clinical Trial Testing Bortezomib in Newly Diagnosed T-Cell Acute Lymphoblastic Leukemia and Lymphoma. J Clin Oncol. 2022 Jul 1;40(19):2106-2118. doi: 10.1200/JCO.21.02678. Epub 2022 Mar 10. PMID 35271306
- [Background] Raetz EA, Rebora P, Conter V, Schrappe M, Devidas M, Escherich G, Imai C, De Moerloose B, Schmiegelow K, Burns MA, Elitzur S, Pieters R, Attarbaschi A, Yeoh A, Pui CH, Stary J, Cario G, Bodmer N, Moorman AV, Buldini B, Vora A, Valsecchi MG. Outcome for Children and Young Adults With T-Cell ALL and Induction Failure in Contemporary Trials. J Clin Oncol. 2023 Nov 10;41(32):5025-5034. doi: 10.1200/JCO.23.00088. Epub 2023 Jul 24. PMID 37487146
- [Background] Polonen P, Di Giacomo D, Seffernick AE, Elsayed A, Kimura S, Benini F, Montefiori LE, Wood BL, Xu J, Chen C, Cheng Z, Newman H, Myers J, Iacobucci I, Li E, Sussman J, Hedges D, Hui Y, Diorio C, Uppuluri L, Frank D, Fan Y, Chang Y, Meshinchi S, Ries R, Shraim R, Li A, Bernt KM, Devidas M, Winter SS, Dunsmore KP, Inaba H, Carroll WL, Ramirez NC, Phillips AH, Kriwacki RW, Yang JJ, Vincent TL, Zhao Y, Ghate PS, Wang J, Reilly C, Zhou X, Sanders MA, Takita J, Kato M, Takasugi N, Chang BH, Press RD, Loh M, Rampersaud E, Raetz E, Hunger SP, Tan K, Chang TC, Wu G, Pounds SB, Mullighan CG, Teachey DT. The genomic basis of childhood T-lineage acute lymphoblastic leukaemia. Nature. 2024 Aug;632(8027):1082-1091. doi: 10.1038/s41586-024-07807-0. Epub 2024 Aug 14. PMID 39143224
- [Background] He Y, Zhang J, Zhang Y, Hu Z, Wang P, Gan W, Xie S, Qian M, Pui CH, Jiang H, Zhu X, Zhang H, Zhang W. Dasatinib-therapy induced sustained remission in a child with refractory TCF7-SPI1 T-cell acute lymphoblastic leukemia. Pediatr Blood Cancer. 2022 Aug;69(8):e29724. doi: 10.1002/pbc.29724. Epub 2022 Apr 20. PMID 35441457
- [Background] Simonin M, Vasseur L, Lengline E, Lhermitte L, Cabannes-Hamy A, Balsat M, Schmidt A, Dourthe ME, Touzart A, Graux C, Grardel N, Cayuela JM, Arnoux I, Gandemer V, Huguet F, Ducassou S, Lheritier V, Chalandon Y, Ifrah N, Dombret H, Macintyre E, Petit A, Rousselot P, Lambert J, Baruchel A, Boissel N, Asnafi V. NGS-based stratification refines the risk stratification in T-ALL and identifies a very-high-risk subgroup of patients. Blood. 2024 Oct 10;144(15):1570-1580. doi: 10.1182/blood.2023023754. PMID 38848537
- [Background] Teachey DT, O'Connor D. How I treat newly diagnosed T-cell acute lymphoblastic leukemia and T-cell lymphoblastic lymphoma in children. Blood. 2020 Jan 16;135(3):159-166. doi: 10.1182/blood.2019001557. PMID 31738819
- [Background] Summers RJ, Teachey DT, Hunger SP. How I treat ETP-ALL in children. Blood. 2025 Jan 2;145(1):43-52. doi: 10.1182/blood.2023023155. PMID 38364183
- [Background] Vora A, Goulden N, Mitchell C, Hancock J, Hough R, Rowntree C, Moorman AV, Wade R. Augmented post-remission therapy for a minimal residual disease-defined high-risk subgroup of children and young people with clinical standard-risk and intermediate-risk acute lymphoblastic leukaemia (UKALL 2003): a randomised controlled trial. Lancet Oncol. 2014 Jul;15(8):809-18. doi: 10.1016/S1470-2045(14)70243-8. Epub 2014 Jun 9. PMID 24924991
- [Background] Schrappe M, Valsecchi MG, Bartram CR, Schrauder A, Panzer-Grumayer R, Moricke A, Parasole R, Zimmermann M, Dworzak M, Buldini B, Reiter A, Basso G, Klingebiel T, Messina C, Ratei R, Cazzaniga G, Koehler R, Locatelli F, Schafer BW, Arico M, Welte K, van Dongen JJ, Gadner H, Biondi A, Conter V. Late MRD response determines relapse risk overall and in subsets of childhood T-cell ALL: results of the AIEOP-BFM-ALL 2000 study. Blood. 2011 Aug 25;118(8):2077-84. doi: 10.1182/blood-2011-03-338707. Epub 2011 Jun 30. PMID 21719599
- [Background] Suo S, Zhao D, Li F, Zhang Y, Rodriguez-Rodriguez S, Nguyen LXT, Ghoda L, Carlesso N, Marcucci G, Zhang B, Jin J. Homoharringtonine inhibits the NOTCH/MYC pathway and exhibits antitumor effects in T-cell acute lymphoblastic leukemia. Blood. 2024 Sep 19;144(12):1343-1347. doi: 10.1182/blood.2023023400. PMID 38968151
- [Background] Chen R, Guo L, Chen Y, Jiang Y, Wierda WG, Plunkett W. Homoharringtonine reduced Mcl-1 expression and induced apoptosis in chronic lymphocytic leukemia. Blood. 2011 Jan 6;117(1):156-64. doi: 10.1182/blood-2010-01-262808. Epub 2010 Oct 22. PMID 20971952
- [Background] Chen XJ, Zhang WN, Chen B, Xi WD, Lu Y, Huang JY, Wang YY, Long J, Wu SF, Zhang YX, Wang S, Li SX, Yin T, Lu M, Xi XD, Li JM, Wang KK, Chen Z, Chen SJ. Homoharringtonine deregulates MYC transcriptional expression by directly binding NF-kappaB repressing factor. Proc Natl Acad Sci U S A. 2019 Feb 5;116(6):2220-2225. doi: 10.1073/pnas.1818539116. Epub 2019 Jan 18. PMID 30659143
- [Background] Lu S, Wang J. Homoharringtonine and omacetaxine for myeloid hematological malignancies. J Hematol Oncol. 2014 Jan 3;7:2. doi: 10.1186/1756-8722-7-2. PMID 24387717
- [Background] Saygin C, Giordano G, Shimamoto K, Eisfelder B, Thomas-Toth A, Venkataraman G, Ananthanarayanan V, Vincent TL, DuVall A, Patel AA, Chen Y, Tan F, Anthony SP, Chen Y, Shen Y, Odenike O, Teachey DT, Kee BL, LaBelle J, Stock W. Dual Targeting of Apoptotic and Signaling Pathways in T-Lineage Acute Lymphoblastic Leukemia. Clin Cancer Res. 2023 Aug 15;29(16):3151-3161. doi: 10.1158/1078-0432.CCR-23-0415. PMID 37363966
- [Background] Shi Y, Beckett MC, Blair HJ, Tirtakusuma R, Nakjang S, Enshaei A, Halsey C, Vormoor J, Heidenreich O, Krippner-Heidenreich A, van Delft FW. Phase II-like murine trial identifies synergy between dexamethasone and dasatinib in T-cell acute lymphoblastic leukemia. Haematologica. 2021 Apr 1;106(4):1056-1066. doi: 10.3324/haematol.2019.241026. PMID 32139432
- [Background] Yoshimura S, Panetta JC, Hu J, Li L, Gocho Y, Du G, Umezawa A, Karol SE, Pui CH, Mullighan CG, Konopleva M, Stock W, Teachey DT, Jain N, Yang JJ. Preclinical pharmacokinetic and pharmacodynamic evaluation of dasatinib and ponatinib for the treatment of T-cell acute lymphoblastic leukemia. Leukemia. 2023 Jun;37(6):1194-1203. doi: 10.1038/s41375-023-01900-5. Epub 2023 Apr 19. PMID 37076694
- [Background] Gocho Y, Liu J, Hu J, Yang W, Dharia NV, Zhang J, Shi H, Du G, John A, Lin TN, Hunt J, Huang X, Ju B, Rowland L, Shi L, Maxwell D, Smart B, Crews KR, Yang W, Hagiwara K, Zhang Y, Roberts K, Wang H, Jabbour E, Stock W, Eisfelder B, Paietta E, Newman S, Roti G, Litzow M, Easton J, Zhang J, Peng J, Chi H, Pounds S, Relling MV, Inaba H, Zhu X, Kornblau S, Pui CH, Konopleva M, Teachey D, Mullighan CG, Stegmaier K, Evans WE, Yu J, Yang JJ. Network-based systems pharmacology reveals heterogeneity in LCK and BCL2 signaling and therapeutic sensitivity of T-cell acute lymphoblastic leukemia. Nat Cancer. 2021 Mar;2(3):284-299. doi: 10.1038/s43018-020-00167-4. Epub 2021 Jan 21. PMID 34151288
- [Background] Lee SHR, Yang W, Gocho Y, John A, Rowland L, Smart B, Williams H, Maxwell D, Hunt J, Yang W, Crews KR, Roberts KG, Jeha S, Cheng C, Karol SE, Relling MV, Rosner GL, Inaba H, Mullighan CG, Pui CH, Evans WE, Yang JJ. Pharmacotypes across the genomic landscape of pediatric acute lymphoblastic leukemia and impact on treatment response. Nat Med. 2023 Jan;29(1):170-179. doi: 10.1038/s41591-022-02112-7. Epub 2023 Jan 5. PMID 36604538
- [Background] Chonghaile TN, Roderick JE, Glenfield C, Ryan J, Sallan SE, Silverman LB, Loh ML, Hunger SP, Wood B, DeAngelo DJ, Stone R, Harris M, Gutierrez A, Kelliher MA, Letai A. Maturation stage of T-cell acute lymphoblastic leukemia determines BCL-2 versus BCL-XL dependence and sensitivity to ABT-199. Cancer Discov. 2014 Sep;4(9):1074-87. doi: 10.1158/2159-8290.CD-14-0353. Epub 2014 Jul 3. PMID 24994123
- [Background] Borah P, Dayal N, Pathak S, Naithani R. Short-course Venetoclax With Standard Chemotherapy Is Effective in Early T-cell Precursor Acute Lymphoblastic Leukemia. J Pediatr Hematol Oncol. 2023 Jul 1;45(5):271-274. doi: 10.1097/MPH.0000000000002672. Epub 2023 Apr 4. PMID 37027330
- [Background] Richard-Carpentier G, Jabbour E, Short NJ, Rausch CR, Savoy JM, Bose P, Yilmaz M, Jain N, Borthakur G, Ohanian M, Alvarado Y, Rytting M, Kebriaei P, Konopleva M, Kantarjian H, Ravandi F. Clinical Experience With Venetoclax Combined With Chemotherapy for Relapsed or Refractory T-Cell Acute Lymphoblastic Leukemia. Clin Lymphoma Myeloma Leuk. 2020 Apr;20(4):212-218. doi: 10.1016/j.clml.2019.09.608. Epub 2019 Sep 30. PMID 32035785
- [Background] Gibson A, Trabal A, McCall D, Khazal S, Toepfer L, Bell DH, Roth M, Mahadeo KM, Nunez C, Short NJ, DiNardo C, Konopleva M, Issa GC, Ravandi F, Jain N, Borthakur G, Kantarjian HM, Jabbour E, Cuglievan B. Venetoclax for Children and Adolescents with Acute Lymphoblastic Leukemia and Lymphoblastic Lymphoma. Cancers (Basel). 2021 Dec 29;14(1):150. doi: 10.3390/cancers14010150. PMID 35008312
- [Background] Davids MS, Letai A. Targeting the B-cell lymphoma/leukemia 2 family in cancer. J Clin Oncol. 2012 Sep 1;30(25):3127-35. doi: 10.1200/JCO.2011.37.0981. Epub 2012 May 29. PMID 22649144
- [Background] Moricke A, Zimmermann M, Valsecchi MG, Stanulla M, Biondi A, Mann G, Locatelli F, Cazzaniga G, Niggli F, Arico M, Bartram CR, Attarbaschi A, Silvestri D, Beier R, Basso G, Ratei R, Kulozik AE, Lo Nigro L, Kremens B, Greiner J, Parasole R, Harbott J, Caruso R, von Stackelberg A, Barisone E, Rossig C, Conter V, Schrappe M. Dexamethasone vs prednisone in induction treatment of pediatric ALL: results of the randomized trial AIEOP-BFM ALL 2000. Blood. 2016 Apr 28;127(17):2101-12. doi: 10.1182/blood-2015-09-670729. Epub 2016 Feb 17. PMID 26888258
- [Background] Campbell M, Kiss C, Zimmermann M, Riccheri C, Kowalczyk J, Felice MS, Kuzmanovic M, Kovacs G, Kosmidis H, Gonzalez A, Bilic E, Castillo L, Kolenova A, Jazbec J, Popa A, Konstantinov D, Kappelmayer J, Szczepanski T, Dworzak M, Buldini B, Gaipa G, Marinov N, Rossi J, Nagy A, Gaspar I, Stary J, Schrappe M. Childhood Acute Lymphoblastic Leukemia: Results of the Randomized Acute Lymphoblastic Leukemia Intercontinental-Berlin-Frankfurt-Munster 2009 Trial. J Clin Oncol. 2023 Jul 1;41(19):3499-3511. doi: 10.1200/JCO.22.01760. Epub 2023 May 4. PMID 37141547
- [Background] Patrick K, Wade R, Goulden N, Mitchell C, Moorman AV, Rowntree C, Jenkinson S, Hough R, Vora A. Outcome for children and young people with Early T-cell precursor acute lymphoblastic leukaemia treated on a contemporary protocol, UKALL 2003. Br J Haematol. 2014 Aug;166(3):421-4. doi: 10.1111/bjh.12882. Epub 2014 Apr 8. PMID 24708207
- [Background] Wood BL, Devidas M, Summers RJ, Chen Z, Asselin B, Rabin KR, Zweidler-McKay PA, Winick NJ, Borowitz MJ, Carroll WL, Raetz EA, Loh ML, Hunger SP, Dunsmore KP, Teachey DT, Winter SS. Prognostic significance of ETP phenotype and minimal residual disease in T-ALL: a Children's Oncology Group study. Blood. 2023 Dec 14;142(24):2069-2078. doi: 10.1182/blood.2023020678. PMID 37556734
- [Background] Morita K, Jain N, Kantarjian H, Takahashi K, Fang H, Konopleva M, El Hussein S, Wang F, Short NJ, Maiti A, Sasaki K, Garcia-Manero G, Konoplev S, Ravandi F, Khoury JD, Jabbour E. Outcome of T-cell acute lymphoblastic leukemia/lymphoma: Focus on near-ETP phenotype and differential impact of nelarabine. Am J Hematol. 2021 May 1;96(5):589-598. doi: 10.1002/ajh.26144. Epub 2021 Mar 18. PMID 33639000
- [Background] Coustan-Smith E, Mullighan CG, Onciu M, Behm FG, Raimondi SC, Pei D, Cheng C, Su X, Rubnitz JE, Basso G, Biondi A, Pui CH, Downing JR, Campana D. Early T-cell precursor leukaemia: a subtype of very high-risk acute lymphoblastic leukaemia. Lancet Oncol. 2009 Feb;10(2):147-56. doi: 10.1016/S1470-2045(08)70314-0. Epub 2009 Jan 13. PMID 19147408
- [Background] Liu Y, Easton J, Shao Y, Maciaszek J, Wang Z, Wilkinson MR, McCastlain K, Edmonson M, Pounds SB, Shi L, Zhou X, Ma X, Sioson E, Li Y, Rusch M, Gupta P, Pei D, Cheng C, Smith MA, Guidry Auvil JM, Gerhard DS, Relling MV, Winick NJ, Carroll AJ, Heerema NA, Raetz E, Devidas M, Willman CL, Harvey RC, Carroll WL, Dunsmore KP, Winter SS, Wood BL, Sorrentino BP, Downing JR, Loh ML, Hunger SP, Zhang J, Mullighan CG. The genomic landscape of pediatric and young adult T-lineage acute lymphoblastic leukemia. Nat Genet. 2017 Aug;49(8):1211-1218. doi: 10.1038/ng.3909. Epub 2017 Jul 3. PMID 28671688
- [Background] Bongiovanni D, Saccomani V, Piovan E. Aberrant Signaling Pathways in T-Cell Acute Lymphoblastic Leukemia. Int J Mol Sci. 2017 Sep 5;18(9):1904. doi: 10.3390/ijms18091904. PMID 28872614
- [Background] Girardi T, Vicente C, Cools J, De Keersmaecker K. The genetics and molecular biology of T-ALL. Blood. 2017 Mar 2;129(9):1113-1123. doi: 10.1182/blood-2016-10-706465. Epub 2017 Jan 23. PMID 28115373
- [Background] Teachey DT, Pui CH. Comparative features and outcomes between paediatric T-cell and B-cell acute lymphoblastic leukaemia. Lancet Oncol. 2019 Mar;20(3):e142-e154. doi: 10.1016/S1470-2045(19)30031-2. PMID 30842058
- [Background] Inaba H, Mullighan CG. Pediatric acute lymphoblastic leukemia. Haematologica. 2020 Nov 1;105(11):2524-2539. doi: 10.3324/haematol.2020.247031. PMID 33054110
- [Background] Hunger SP, Mullighan CG. Acute Lymphoblastic Leukemia in Children. N Engl J Med. 2015 Oct 15;373(16):1541-52. doi: 10.1056/NEJMra1400972. No abstract available. PMID 26465987
- Available data/document: Individual Participant Data Set: CCCG-ALL — http://cccg.nipher.com/cccg/ — CCCG-ALL-2025 DATASET